CLINICAL TRIAL: NCT00704938
Title: Phase II Study of Metastatic Cancer That Overexpresses p53 Using Lymphodepleting Conditioning Followed by Infusion of Anti-P53 TCR-Gene Engineered Lymphocytes and Dendritic Cell Vaccination
Brief Title: Gene-Modified Lymphocytes, High-Dose Aldesleukin, and Vaccine Therapy in Treating Patients With Progressive or Recurrent Metastatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to withdrawal of support from our collaborator.
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080155; NCI-08-C-0155; NCI-P07215
Record Dates: First submitted 2008-06-24; First posted 2008-06-25 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-09

CONDITIONS: Kidney Cancer; Melanoma (Skin); Unspecified Adult Solid Tumor, Protocol Specific
Keywords: recurrent renal cell cancer; stage IV renal cell cancer; recurrent melanoma; stage IV melanoma; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — aldesleukin; Filgrastim; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anti-p53 TCR PBL + DC + IL-2: Melanoma/RCC (Experimental): Patients with melanoma and renal cell cancer will receive anti-p53 T cell receptor (TCR) peripheral blood lymphocytes (PBL) + dendritic cells (DC) + interleukin-2 (IL-2)
  Interventions: Biological: aldesleukin; Biological: anti-p53 T-cell receptor-transduced peripheral blood lymphocytes; Biological: autologous dendritic cell-adenovirus p53 vaccine; Biological: filgrastim; Drug: cyclophosphamide; Drug: fludarabine phosphate
- anti-p53 TCR PBL + DC + IL-2: Other histology (Experimental): Patients with other histologies, such as breast cancer, will receive anti-p53 T cell receptor (TCR) peripheral blood lymphocytes (PBL) + dendritic cells (DC) + interleukin-2 (IL-2)
  Interventions: Biological: aldesleukin; Biological: anti-p53 T-cell receptor-transduced peripheral blood lymphocytes; Biological: autologous dendritic cell-adenovirus p53 vaccine; Biological: filgrastim; Drug: cyclophosphamide; Drug: fludarabine phosphate

INTERVENTIONS:
Biological: aldesleukin — Intravenous (IV) aldesleukin 720,000 IU/kg every 8 hours for a maximum of 15 doses.
  Other Names: Proleukin
Biological: anti-p53 T-cell receptor-transduced peripheral blood lymphocytes — Intravenous (IV) anti-p53 TCR transduced PBL will be administered at a a dose of 1 x 10^8 cells to 5 x 10^10 cells.
Biological: autologous dendritic cell-adenovirus p53 vaccine — Ad-p53 DC vaccine, up to 2 x 10^8 ad-p53 DCs per dose will be administered subcutaneously, divided into 4 injections, one into each of the 4 extremities. Ad-p53 DCs will be administered subcutaneously on day 7 (± 2 days), day 14 (between day 14 and day 18), and day 28 (between day 25 and day 42) post T cell infusion.
Biological: filgrastim — subcutaneously at a dose of 5 mcg/kg/day (not to exceed 300 mcg/day).
  Other Names: growth colony stimulating factor (GCSF)
Drug: cyclophosphamide — 60mg/kg/day (Days-7,-6)
  Other Names: Cytoxan
Drug: fludarabine phosphate — 25mg/m^2 (Days -5, -4, -3, -2, and -1)
  Other Names: Fludara

SUMMARY:
RATIONALE: Gene-modified lymphocytes may stimulate the immune system in different ways and stop tumor cells from growing. High-dose aldesleukin may stimulate lymphocytes to kill tumor cells. Vaccines made from a gene modified virus and a person's dendritic cells may help the body build an effective immune response to kill tumor cells. Giving gene-modified lymphocytes together with high-dose aldesleukin and vaccine therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gene-modified lymphocytes together with high-dose aldesleukin and vaccine therapy works in treating patients with progressive or recurrent metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if the administration of anti-p53 T-cell receptor (TCR) gene-engineered peripheral blood lymphocytes, high-dose aldesleukin, and adenovirus p53 dendritic cell (DC) vaccine after a nonmyeloablative, but lymphoid-depleting, preparative regimen will result in clinical tumor regression in patients with metastatic cancer that overexpresses p53.

Secondary

* Determine the in vivo survival of T-cell receptor (TCR) gene-engineered cells.
* Determine the ability of a dendritic cell (DC) vaccine to restimulate TCR gene-engineered cells in vivo.
* Determine the toxicity profile of this treatment regimen.

OUTLINE: Patients are stratified according to type of metastatic cancer (melanoma or renal cell cancer vs all other cancers).

* Peripheral blood mononuclear cell (PBMC) collection: Patients undergo PBMC collection via leukapheresis for the generation of the adenovirus p53 dendritic cell vaccine as well as anti-p53 T-cell receptor (TCR) gene-engineered peripheral blood lymphocytes.
* Nonmyeloablative lymphocyte-depleting preparative regimen: Patients receive cyclophosphamide intravenously (IV) over 1 hour on days -7 and -6 and fludarabine phosphate IV over 30 minutes on days -5 to -1.
* Peripheral blood lymphocyte infusion: Patients receive anti-p53 TCR gene-engineered peripheral blood lymphocytes IV over 20-30 minutes on day 0. Patients receive filgrastim (growth colony stimulating factor (G-CSF)) subcutaneously (SC) once daily beginning on day 1 or 2 and continuing until blood counts recover.
* High-dose aldesleukin: Patients receive high-dose aldesleukin IV over 15 minutes three times daily on days 0-4 for up to 15 doses.
* Dendritic cell vaccine: Patients receive adenovirus p53 dendritic cell vaccine SC on days 0, 7, 14, and 28.

Patients may receive one re-treatment course as above (nonmyeloablative preparative regimen, peripheral blood lymphocyte infusion, high-dose aldesleukin, and dendritic cell vaccinations) beginning 6-8 weeks after the last dose of high-dose aldesleukin.

After completion of study treatment, patients are followed periodically for up to 15 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic cancer
* Tumor overexpresses p53 as assessed by immunohistochemistry (i.e., ≥ 5% tumor cells stain positive for p53)

  * Biopsy must be available to evaluate p53 expression
* Human leukocyte antigens 0201 (HLA-A*0201) positive
* Progressive or recurrent disease after prior standard therapy for metastatic disease

  * Patients with melanoma or renal cell cancer must have previously received aldesleukin
  * Patients with other histologies, not including hematologic malignancies, must have previously received first-line and second-line or higher systemic standard therapy (or effective salvage chemotherapy regimens)

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy > 3 months
* Absolute neutrophil count > 1,000/mm^3
* White blood cell (WBC) > 3,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 8.0 g/dL
* Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 2.5 times upper limit of normal
* Serum creatinine ≤ 1.6 mg/dL
* Total bilirubin ≤ 2.0 mg/dL (< 3.0 mg/dL in patients with Gilbert's syndrome)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 months after completion of study treatment
* Patients who have previously received ipilimumab or ticilimumab must have a normal colonoscopy with normal colonic biopsies
* Human immunodeficiency virus (HIV) antibody negative
* Hepatitis B antigen and hepatitis C antibody negative (unless antigen negative)
* No primary immunodeficiency (e.g., severe combined immunodeficiency disease)
* No active systemic infections
* No history of severe immediate hypersensitivity reaction to any of the agents used in this study
* No coagulation disorders
* No myocardial infarction or cardiac arrhythmias
* No history of coronary revascularization
* No obstructive or restrictive pulmonary disease
* No contraindications for high-dose aldesleukin administration
* Left ventricular ejection fraction (LVEF) ≥ 45% in patients meeting any of the following criteria:

  * History of ischemic heart disease,
  * chest pain,
  * or clinically significant atrial and/or ventricular arrhythmias including, but not limited to, atrial fibrillation,
  * ventricular tachycardia,
  * or second- or third-degree heart block
  * At least 60 years of age
* Forced expiratory volume 1 (FEV_1) > 60% predicted in patients meeting any of the following criteria:

  * Prolonged history of cigarette smoking (> 20 pack/year within the past 2 years)
  * Symptoms of respiratory dysfunction
* No other major medical illness of the cardiovascular,

  * respiratory,
  * or immune system

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* More than 4 weeks since prior and no concurrent systemic steroid therapy
* More than 4 weeks since other prior systemic therapy
* More than 6 weeks since prior ipilimumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Principal Investigator — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Anti-p53 TCR PBL + DC + IL-2: Other Histology: Patients with other histologies will receive anti-p53 T cell receptor (TCR) peripheral blood lymphocytes (PBL) + dendritic cells (DC) + interleukin-2 (IL-2)
Period: Overall Study
Arm/Group | Anti-p53 TCR PBL + DC + IL-2: Melanoma/RCC | Anti-p53 TCR PBL + DC + IL-2: Other Histology
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-p53 TCR PBL + DC + IL-2: Melanoma/RCC | Anti-p53 TCR PBL + DC + IL-2: Other Histology | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (13.4) | 58.0 | 47.25 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response (Complete Response + Partial Response)
Description: Clinical response is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is disappearance of all lesions. Partial response is a 30% decrease in the sum of the longest diameter (LD) of target lesions.
Time Frame: 5 months
Measure: Number; unit: Participants
Arm/Group | Anti-p53 TCR PBL + DC + IL-2: Melanoma/RCC | Anti-p53 TCR PBL + DC + IL-2: Other Histology
Number analyzed (Participants) | 2 | 1
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse events module.
Time Frame: 5 months
Measure: Number; unit: Participants
Arm/Group | Anti-p53 TCR PBL + DC + IL-2: Melanoma/RCC | Anti-p53 TCR PBL + DC + IL-2: Other Histology
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Anti-p53 TCR PBL + DC + IL-2: Melanoma/RCC | Anti-p53 TCR PBL + DC + IL-2: Other Histology
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-p53 TCR PBL + DC + IL-2: Melanoma/RCC (N=2) | Anti-p53 TCR PBL + DC + IL-2: Other Histology (N=1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Leukocyte count decreased (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
lymphocyte count decreased (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Optic nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Nervous system disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Low urine output (Renal and urinary disorders) | 1 (2) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated prior to completing accrual due to the withdrawal of support from our collaborator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No